CLINICAL TRIAL: NCT05004701
Title: Impact of the Lockdown Due to the COVID Pandemic in French Wilson's Disease Patients
Acronym: WILL-Ecco
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: APS_2020_17
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Wilson's Disease and COVID-19
MeSH Terms: conditions — Hepatolenticular Degeneration; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Wilson's disease is a rare genetic disorder that causes copper to build up in the body. This overload is initially localized in the liver and the brain, but can spread throughout the body and cause systemic damage if copper chelation or zinc salt therapy is not implemented quickly. Treatment should be taken daily and continued all the lifelong.

Patients usually have a follow-up (clinical examination, ultrasound of the liver, blood and urine samples) every six months in the maintenance phase of the disease and more frequently in the event of destabilization of the disease which requires adaptation of the doses of treatment or when initiating treatment. Some patients also benefit from regular psychological follow-up and patients with a disabling neurological form may have physiotherapy, and speech therapy. The Covid 19 pandemic has imposed the lockdown of the entire population, including patients with Wilson's disease. The non-urgent care of these patients was therefore suspended. Medical consultations and paramedical care (physiotherapy, speech therapy, psychologist, etc.) have been postponed. Only very urgent hospitalizations in the event of imbalance of their illness with life-threatening risk were maintained.

Wilson's disease patients could in this situation be particularly anxious and present disturbances of their quality of life. The psychiatric consequences could not be limited to the current period but also concern long-term patients, in particular if there is a worsening of the disease. The consequences of inactivity and the end of specific treatments (physiotherapy and speech therapy) could also be sources of aggravation. The behavioral and cognitive characteristics of the disease and the major difficulties in adherence to treatment already observed in this chronic disease, may suggest a repercussion of the pandemic in this population.

The consequences of the COVID pandemic in these fragile patients with a rare disease must be assessed. It will be important to look at the consequences of the lockdown on the adherence to treatment and on the course of the disease.

DETAILED DESCRIPTION:
During the lockdown period, the first part of a detailed questionnaire is proposed to Wilson's disease patients. The second part of the questionnaire will be carried out away from the lockdown This is an observational, French multicenter study, of an uncontrolled cohort of Wilsonian patients followed by doctors from the Wilson national reference centers

Intervention 1:

Other: Questionnaires The questionnaires are WHOQOL-BREF (quality of life) Compliance questionnaire with a Visual Analog Scale (VAS) from 0 to 100 Hospital Anxiety and Depression scale (HAD)

ELIGIBILITY:
Inclusion Criteria:

* Wilson's disease patient
* Patient over 12 years of age
* Patient followed by doctors from the Wilson national reference centers (Paris, Lyon, Toulouse, Besançon, Bordeaux, Rennes, Marseilles, Tours, Lille )
* Patients hospitalized or seen in outpatient consultation (or teleconsultation) during the first confinement and at the end of the last one
* Non-opposition of participation in the study and for minor patient non-opposition of one of the two holders of the exercise of parental authority

Exclusion criteria :

* Patient subject to a legal protection (tutorship)
* Patient or patient representative not wishing to answer questions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Wilson's disease followed by doctors from the Wilson national reference centers between the first confinement due to COVID and the end of the last lockdown
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Quality of life was measured using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire | 6 months
  To describe the quality of life of Wilsonian patients during the COVID lockdown and at short and long term after it. Quality of life was measured using the WHOQOL-BREF questionnaire The WHOQOL-BREF is a self-administered questionnaire comprising 26 questions on the individual's perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
  Thethe World Health Organization Quality of Life-BREF ( WHOQOL-BREF ) covers four domains each with specific facets

CONTACTS AND LOCATIONS:
Overall Officials: Aurélia Poujois, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A De Rothschild, Paris, France